CLINICAL TRIAL: NCT05493436
Title: The Influence of Obesity to Esophageal Reflux Severity Measured by pH-Metri Impedans on Gastroesophageal Reflux Disease Patients
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ari Fahrial Syam, Clinical Professor, Staff of Gastroenterology Division, Department of Internal Medicine, Indonesia University
Other Study IDs: IndonesiaSatu
Record Dates: First submitted 2020-08-12; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Disorder of Upper Esophageal Sphincter

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normoweight: GERD patient with normoweight was evaluating by MII pH-meter
  Interventions: Diagnostic Test: MII pH-meter
- obesity: GERD patient with obesity was evaluating by MII pH-meter
  Interventions: Diagnostic Test: MII pH-meter

INTERVENTIONS:
Diagnostic Test: MII pH-meter — using multichannel impedance pH-meter

SUMMARY:
To see a more convincing relationship between increased body mass index and the severity of esophageal reflux in GERD patients, GERD diagnosis should be performed with greater precision or precision. From the available data, it appears that no studies in Indonesia have correlated the body mass index with the severity of esophageal reflux events measured by multical intraluminal intraluminal pH-metric in patients with GERD due to the invasive nature of the test. Therefore, research needs to be done to assess the effect of increased body mass index on the severity of esophageal reflux as measured by multical intraluminal impedance pH-metric in GERD patients.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) prevalence is increasing worldwide. It is known that GERD correlates with obesity. In order to see further association between obesity and severity degree of esophageal reflux, GERD must be diagnosed with greater precision and accuracy. Therefore, study to see the impact of obesity in esophageal reflux severity measured by multicanal intraluminal impedance pH-meter (MII-pH) in GERD patient is compulsory.

The objective of this study is to explain the impact of obesity on severity of esophageal reflux in GERD patient measured by DeMeester score, hiatal hernia incidence, and the prolongation of acid exposure time in GERD patient.

This cross-sectional study recruited patients from Gastroenterology Clinic, Internal Medicine Department Cipto Mangunkusumo Hospital during May-August 2017. Patient with normal and obese body mass index (BMI) suspected having GERD were surveyed using GERDQ to diagnose GERD in these patients. Upper gastrointestinal endoscopy were performed to see hiatal hernia. All patients recruited underwent MII-pH examination to measure DeMeester score and acid exposure time. Results were analyzed using bivariat analysis.

ELIGIBILITY:
Inclusion Criteria:

1. GERD patients diagnosed by GerdQ
2. Adult patient age 18-60 years
3. Patients with nutritional status based on normal BMI (18.5-24.9) and obesity (≥30)
4. Willing to participate in research and sign informed consent

Exclusion Criteria:

1. At the endoscopic examination found Barrett's esophagus, peptic ulcer, severe gastritis, severe NSAID gastropathy, hemorrhage (melenae), gastric cancer, esophageal cancer
2. MII-pH check failed to install
3. Patients are not cooperative
4. Patients with acute psychiatric disorders
5. Patients with severe heart trouble, persistent asthma patients, decompensated liver cirrhosis and chronic renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with GERD
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Composite pH score/DeMesster Score | January 2017 - October 2017
  Participants underwent multichannel intraluminal impedance pH-meter (MII-pH) monitoring for quantification of the DeMeester score and acid exposure time

SECONDARY OUTCOMES:
Acid exposure time | January 2017 - October 2017
  Percent of acid exposure time (AET) at pH < 4 for each study groups
Incidence of Hiatal Hernia | January 2017 - October 2017
  Incidence of hiatal hernia is measured for each group
Incidence of Erosive Esophagitis | January 2017 - October 2017
  Incidence of erosive esophagitis is measured for each group

CONTACTS AND LOCATIONS:
Locations (1):
- RSCM, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05493436/Prot_SAP_ICF_000.pdf